CLINICAL TRIAL: NCT04971317
Title: The Influence of Simple, Low-Cost Chemistry Intervention Videos: A Randomized Trial of Children's Preferences for Sugar-Sweetened Beverages"
Brief Title: The Influence of Simple, Low-Cost Chemistry Intervention Videos: A Randomized Trial of Children's Preferences for Sugar-Sweetened Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-00048
Record Dates: First submitted 2021-07-14; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Type 2 Diabetes; Dental Caries
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Dental Caries | interventions — Sugar-Sweetened Beverages; SSB protein, human; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sugar-Sweetened Beverage (SSB) Video (Experimental)
  Interventions: Behavioral: Sugar-Sweetened Beverage (SSB) Video
- Water Video (Experimental)
  Interventions: Behavioral: Water Video
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Sugar-Sweetened Beverage (SSB) Video — Participants will watch a video showing the decay of an egg in various SSBs (Coca-Cola, Sprite, Gatorade, and apple juice), followed by the evaporation of these beverages over a heat source, revealing their sugar content.
  Arms: Sugar-Sweetened Beverage (SSB) Video
Behavioral: Water Video — Participants will watch a video showing an egg maintaining its shell in water, followed by the evaporation of water.
  Arms: Water Video
Behavioral: Control — Participants will watch a video of an egg maintaining its shell in rubbing alcohol, followed by the evaporation of rubbing alcohol.
  Arms: Control

SUMMARY:
Sugar-sweetened beverage (SSB) consumption is associated with the development of obesity, type 2 diabetes, and dental caries. The current study attempts to explore whether an educational, science-based intervention is able to produce a measurable negative change in preferences for sugar-sweetened beverages, as well as initiate plans to reduce future SSB consumption in 12-year old children. In the first condition (SSB Intervention), participants will watch a video showing the decay of an egg in various SSBs (Coca-Cola, Sprite, Gatorade, and apple juice), followed by the evaporation of these beverages over a heat source, revealing their sugar content. In the second condition (Water Intervention), participants will watch a video showing an egg maintaining its shell in water, followed by the evaporation of water. In the third condition (Control), participants will watch a video of an egg maintaining its shell in rubbing alcohol, followed by the evaporation of rubbing alcohol. Before and after watching their assigned video, participants will complete survey questions to assess self-reported: SSB consumption intentions, attitudes toward SSBs, and health perceptions of SSBs. Therefore, the aims of this study are to (1) quantify changes in SSB consumption intentions, attitudes towards SSBs, and health perceptions of SSBs from pre-video to post-video, (2) establish the effectiveness of the SSB Intervention and Water Intervention over the control, (3) establish the effectiveness of the SSB Intervention over the Water Intervention, (4) determine the efficacy of incorporating scientific evidence in a public health intervention, and (5) make recommendations for the future application of the method employed in this intervention to future public health campaigns.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit a nationally representative sample of participants through the subdivision of Qualtrics, Qualtrics Panel. Participants must be 12 years old and English speaking.

Exclusion Criteria:

* Any participant that is not 12 years old or does not speak English will be excluded from participation.

Ages: 12 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 326 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Frequency of SSB Consumption | 30 days
  Measurement of how often participants consume various SSBs using the following questions: 1) During the past 30 days, how often did you drink regular soda or pop that contains sugar (such as Coca-Cola, Pepsi, Sprite, Mountain Dew, 7Up, Dr. Pepper, Ginger Ale, Fanta, etc.)? Do not include diet soda or diet pop. 2) During the past 30 days, how often did you drink sports drinks (such as Gatorade, Powerade, Vitamin Water, etc.)? Do not include diet drinks or artificially sweetened drinks. 3) During the past 30 days, how often did you drink sugar-sweetened fruit drinks (such as Kool-aid, lemonade, cranberry juice, etc.)? Do not include 100% fruit juice.
  *Questions have been adapted from the BRFSS Sugar Sweetened Beverage Optional Module
Attitudes towards SSBs | 30 days
  Attitudes to SSBs will be assessed using the following questions measured on a 7-point likert scale: 1) I feel positive toward soda or pop/I feel negative toward soda or pop (such as Coca-Cola, Pepsi, Sprite, Mountain Dew, 7Up, Dr. Pepper, Ginger Ale, Fanta, etc.). Do not include diet soda or diet pop. 2) I feel positive toward sports drinks/I feel negative toward sports drinks (such as Gatorade, Powerade, Vitamin Water, etc.)? Do not include diet drinks or artificially sweetened drinks. 3) I feel positive toward sugar-sweetened fruit drinks/I feel negative toward sugar-sweetened fruit drinks (such as Kool-aid, lemonade, cranberry juice, etc.). Do not include 100% fruit juice.
Health Perceptions of SSBs | 30 days
  Response to SSBs will be assessed using the following questions measured on a 7-point likert scale: 1) I think that soda or pop (such as Coca-Cola, Pepsi, Sprite, Mountain Dew, 7Up, Dr. Pepper, Ginger Ale, Fanta, etc.) is healthy/unhealthy. Do not include diet soda or diet pop. 2) I think that sports drinks (such as Gatorade, Powerade, Vitamin Water, etc.) are healthy/unhealthy. Do not include diet drinks or artificially sweetened drinks. 3) I think that fruit drinks (such as Kool-aid, lemonade, cranberry juice, etc.) are healthy/unhealthy. Do not include 100% fruit juice.
Plans for Future SSB Consumption Post-Intervention or Post-Control | 30 days
  Measurement of how often participants plan to consume various SSBs using the following questions: 1) During the next 30 days, how often do you plan on drinking regular soda or pop that contains sugar (such as Coca-Cola, Pepsi, Sprite, Mountain Dew, 7Up, Dr. Pepper, Ginger Ale, Fanta, etc.)? Do not include diet soda or diet pop. 2) During the next 30 days, how often do you plan on drinking sports drinks (such as Gatorade, Powerade, Vitamin Water, etc.)? Do not include diet drinks or artificially sweetened drinks. 3) During the next 30 days, how often do you plan on drinking sugar-sweetened fruit drinks (such as Kool-aid, lemonade, cranberry juice, etc.)? Do not include 100% fruit juice.
Attitudes towards SSBs Post-Intervention or Post-Control | 30 days
  Response to SSBs will be assessed using the following questions measured on a 7-point likert scale: 1) I feel positive toward soda or pop/I feel negative toward soda or pop (such as Coca-Cola, Pepsi, Sprite, Mountain Dew, 7Up, Dr. Pepper, Ginger Ale, Fanta, etc.). Do not include diet soda or diet pop. 2) I feel positive toward sports drinks/I feel negative toward sports drinks (such as Gatorade, Powerade, Vitamin Water, etc.)? Do not include diet drinks or artificially sweetened drinks. 3) I feel positive toward sugar-sweetened fruit drinks/I feel negative toward sugar-sweetened fruit drinks (such as Kool-aid, lemonade, cranberry juice, etc.). Do not include 100% fruit juice.
Health Perceptions of SSBs Post-Intervention or Post-Control | 30 days
  Response to SSBs will be assessed using the following questions measured on a 7-point likert scale: 1) I think that soda or pop (such as Coca-Cola, Pepsi, Sprite, Mountain Dew, 7Up, Dr. Pepper, Ginger Ale, Fanta, etc.) is healthy/unhealthy. Do not include diet soda or diet pop. 2) I think that sports drinks (such as Gatorade, Powerade, Vitamin Water, etc.) are healthy/unhealthy. Do not include diet drinks or artificially sweetened drinks. 3) I think that fruit drinks (such as Kool-aid, lemonade, cranberry juice, etc.) are healthy/unhealthy. Do not include 100% fruit juice.

CONTACTS AND LOCATIONS:
Overall Officials: Marie A Bragg, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to the PI. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP